# LIVE-C-FREE (LIVEr transplant for hepatitis C: recurrence FREE)

Early and late treatment of Hepatitis C with Sofosbuvir/Ledipasvir in Liver Transplant Recipients

## **Study Chair:**

Derek A. DuBay, MD
Associate Professor of Surgery
Chief, Division of Transplant Surgery
Medical University of South Carolina

**Supported by:** 

Gilead Sciences IN-US-337-1830

Study Intervention Provided by: Gilead Sciences

**Sponsor of Study:** Derek DuBay/MUSC

ClinicalTrials.gov NCT02631772

Protocol Version 6
Protocol Version Date: March 7, 2017

(Any modification to the protocol should be annotated on the coversheet or in an appendix. The annotation should note the exact words that are changed, the location in the protocol, the date the modification was approved by the Executive Committee, and the date it became effective.)

# TABLE OF CONTENTS

| 1. STUDY OBJECTIVES | 4 |
|---------------------------------------------------------|----|
| 1.1 Primary Objective | 4 |
| 1.2 SECONDARY OBJECTIVES | 4 |
| 2. BACKGROUND | 4 |
| 2.1 Rationale | 4 |
| 2.2 SUPPORTING DATA | 5 |
| 3. STUDY DESIGN | 6 |
| 4. SELECTION AND ENROLLMENT OF SUBJECTS | 7 |
| 4.1 Inclusion Criteria | 7 |
| 4.2 Exclusion Criteria | 7 |
| 4.3 STUDY ENROLLMENT PROCEDURES | 8 |
| 5. STUDY INTERVENTIONS | 10 |
| 5.1 Interventions, Administration, and Duration | 10 |
| 5.2 Prohibited Interventions | 12 |
| 5.3 ADHERENCE ASSESSMENT | 13 |
| 6. CLINICAL AND LABORATORY EVALUATIONS | 14 |
| 6.1 SCHEDULE OF EVALUATIONS | 14 |
| 6.2 Timing of Evaluations | 14 |
| 7. MANAGEMENT OF COMMON OR EXPECTED ADVERSE EXPERIENCES | 16 |
| 8. CRITERIA FOR INTERVENTION DISCONTINUATION | 23 |
| 9. STATISTICAL CONSIDERATIONS | |
| 9.1 General Design Issues | 24 |
| 9 2 Outcomes | 25 |

| | version 6 |
|---|---|
| 9.3 SAMPLE SIZE ESTIMATION FOR THE PRIMARY OUTCOME | 25 |
| 9.4 STATISTICAL EVALUATION OF PRIMARY ENDPOINT | 25 |
| 9.5 MISSING DATA AND IMPUTATION METHODS ERR | OR! BOOKMARK NOT DEFINED. |
| 9.6 SECONDARY ENDPOINTS ERRO | OR! BOOKMARK NOT DEFINED. |
| 9.7 SAFETY ANALYSIS | 26 |
| 10. DATA COLLECTION, SITE MONITORING, ADVERSE | EVENT REPORTING 27 |
| 10.1 Data Processing | 27 |
| 10.2 Data Security and Confidentiality | 28 |
| 10.3 Data Quality Assurance | 28 |
| 10.4 Adverse Experience Reporting | 29 |
| 11. HUMAN SUBJECTS | 30 |
| 11.1 INSTITUTIONAL REVIEW BOARD (IRB) REVIEW AND INFORM | MED CONSENT 30 |
| 11.2 STUDY MODIFICATION/DISCONTINUATION | 30 |
| 12. PUBLICATION OF RESEARCH FINDINGS | 30 |
| 13. REFERENCES | 31 |
| APPENDIX I | 32 |
| APPENDIX II | 33 |

#### 1. STUDY OBJECTIVES

## 1.1 Primary Objective

LDV/SOF for 12 weeks will have an equivalent SVR12 compared to LDV/SOF+ribavirin for 12 weeks, both initiated after liver transplant.

## 1.2 Secondary Objectives

Secondary objectives include the emergence and effect of NS5A and NS5B viral substitutions at baseline and in the event of relapse.

### 2. BACKGROUND

#### 2.1 Rationale

Therapeutic response rates for the treatment of recurrent hepatitis C virus (HCV) after liver transplant have historically lagged behind non-transplant patients (1). While the latest studies in HCV therapy with new direct-acting antivirals (DAA) have drastically improved sustained virologic response rates (SVR) in non-transplant patients, HCV is still the most common cause of end stage liver disease (ESLD) leading to liver transplant (2,3,4,5). Although the DAAs have shown efficacy in recurrent HCV post-transplant, this is with late treatment, since preemptive therapy has not shown benefit with previous agents (6,7). An attempt at preventing recurrence by clearing the virus with SOF and RBV prior to transplant has shown encouraging preliminary results in patients who had HCV RNA undetectability for  $\geq$  30 days, however this was in well-compensated cirrhotics (CTP  $\leq$  7) with concomitant HCC (8). Due to the poor tolerability of RBV in patients with more advanced cirrhosis, it is unknown if this regimen would have external validity to the overall HCV population awaiting liver transplant. Also complicating the reproducibility of this data is the unpredictable timing of liver transplant surgery.

Preliminary results of the ongoing SOLAR-1 study have shown excellent sustained virologic response (SVR) rates with 12 weeks of therapy both pre and post-transplant, when utilizing a regimen of LDV/SOF and RBV (9). However, this is with a regimen that includes an antiviral with poor tolerability post-transplant, ribavirin.

The predominant remaining questions for post-transplant treatment of HCV in the DAA era are whether a ribavirin-free regimen is possible and whether pre-emptive treatment is now a potential option to prevent long-term damage to the allograft.

Version 6

These questions require formal testing in a clinical trial conducted in transplant centers.

# 2.2 Supporting Data

SOLAR-1 – Phase III randomized, open-label study including post-transplant (Cohort B) (ongoing)



## a. Results

## Post-transplant F0-F3, CPT A/B/C (cohort B)

- i. N=223, 12 vs 24 wks of LDV/SOF+riba (weight-based in F0-F3 and CPT A, 600mg titrated up in CPT B and C)
- ii. Median time since transplant 2.9-8.1 yrs depending on arm
- iii. SVR rate
  - 1. F0-F3 96-98% (N=111)
  - 2. CPT A 96-96% (N=51)
  - 3. CPT B 85-83% (N=44)
  - 4. CPT C (N=8) (only 9 pts in this arm, 1 has not reached SVR endpoint timeframe) 60-67%

# Risks of therapy

| | HARVONI 8 weeks | HARVONI 12 weeks | HARVONI 24 weeks |
|----------------------|-----------------|------------------|------------------|
| | N=215 | N=539 | N=326 |
| Fatigue | 16% | 13% | 18% |
| Headache | 11% | 14% | 17% |
| Nausea | 6% | 7% | 9% |
| Diarrhea | 4% | 3% | 7% |
| Insomnia | 3% | 5% | 6% |
| Bilirubin elevations | 3% | <1% | 2% |
| 1.5x ULN | | | |
| Lipase elevations | <1% | 2% | 3% |
| 3x ULN | | | |

# 3. STUDY DESIGN

Multi-center, prospective, randomized, open-label, pilot study

ARM 1: LDV/SOF x 12 weeks

ARM 2: LDV/SOF + RBV x 12 weeks

# **Number subjects**:

Multi-center

50 subjects, with 25 subjects in each arm

### 4. SELECTION AND ENROLLMENT OF SUBJECTS

#### 4.1 Inclusion Criteria

- a. At least 18 years of age
- b. Signed informed consent
- c. History of HCV genotype 1 or 4
- d. No clinically significant abnormalities or changes on EKG
- e. Randomization post orthotopic liver transplant
- f. Detectable HCV RNA at baseline
- g. Creatinine Clearance of at least 40ml/min using the Cockcroft Gault equation
- h. Negative pregnancy test for female subjects of child bearing potential within 48 hours of randomization

Subjects of reproductive potential agree to use (or have their partner use) two effective contraception methods through 6 weeks following completion of intervention. Subjects who are not of reproductive potential, not sexually active, whose current partner(s) is not of reproductive potential, or whose sexual activity is exclusively homosexual are eligible without requiring the use of contraception.

### 4.2 Exclusion Criteria

- a. Pregnant or nursing female, or male with a pregnant female partner
- b. A condition or disorder that, in the opinion of the investigator, may adversely affect the outcome of the study or the safety of the subject
- c. Stomach disorder that could interfere with the absorption of study drug
- d. Co-infected with HBV or HIV
- e. Allergic to sofosbuvir or ledipasvir
- f. History of completed treatment with a Nonstructural Protein 5A (NS5a) inhibitor

- g. Participation in a clinical study with an investigational drug or biologic within 30 days of randomization
- h. Fibrosing cholestatic hepatitis
- i. Amiodarone use within 6 months of randomization
- j. Unwilling/unable to stop taking any of the prohibited medications (Section 5.2)
- k. Total bilirubin >10mg/dL
- l. Alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase (ALP)  $\geq 10x$  ULN
- m. Serum sodium < 125mmol/L
- n. Platelet count of  $\leq 30 \text{ k/mm}^3$
- o. Hemoglobin < 10g/dL
- p. Allergic to or intolerant of ribavirin
- q. Within 1 year of transplant AND history of Hepatocellular Carcinoma (HCC) with tumor burden outside of the Milan Criteria (See Appendix II) prior to transplant
- r. History of significant or unstable cardiac disease
- s. Recipients of an allograft from a donor that was infected with HCV with an unknown genotype or non-genotype 1 or 4 unless the recipient is demonstrated to have only genotype 1 or 4 HCV replication post-transplant
- t. Childs Turcotte Pugh (CTP) B or C

### 4.3 Study Enrollment Procedures

- 4.3.1 Subject Identification/Recruitment: Members of the research team will identify potentially eligible patients who are undergoing liver transplantation or have previously undergone liver transplantation that are infected with Hepatitis C. An initial evaluation of existing patient information may be performed to determine potential eligibility. This initial review may be performed prior to consent; however no protocol driven tests or procedures may be performed until signed informed consent has been obtained.
- 4.3.2 Informed Consent: Authorized personnel will approach patients to explain the study and offer the opportunity to participate in the study. The personnel who will obtain

Version 6

consent will have completed Human Subjects Protection Training. This research study will be explained in lay terms to each potential research participant. In compliance with the informed consent process outlined in CFR Title 21 Part 50, the authorized personnel will conduct a face-to-face meeting with the study candidate to review all of the required elements of informed consent. The potential study participant will sign an informed consent form before undergoing any screening study procedures. The original consent form will be kept with the subject's file in the office. A copy of the consent will be given to the patient and another copy will be put in his/her chart. At the time of consent, patients will be assured that their care will not be affected in any way if they choose not to participate in the study. Patients will also be reminded that it is their right to withdraw their participation in the study at any time.

4.3.3 Enrollment: Patients who give informed consent to study participation will go on to complete baseline procedures necessary to determine eligibility for randomization. Once deemed eligible for the study according to the inclusion/exclusion criteria, the patient will be enrolled as study subject in the WebDCU<sup>TM</sup> clinical trial management system (CTMS). Information to be entered upon enrollment includes demographic information and date of transplant surgery. Enrolled subjects will be randomized to one of the treatment arms. The study team will receive the randomization assignment from WebDCU<sup>TM</sup>.

### 5. STUDY INTERVENTIONS

### 5.1 Interventions, Administration, and Duration

# i. SOF/LDV administration

At the time of randomization, all subjects will be initiated on SOF/LDV 400mg/90mg enterally daily either with food or on an empty stomach. This medication will be administered predominantly outpatient, although it may be started or continued on both general hospital floors as well as the ICU. The medication will be continued for 12 weeks in both arms.

## ii. Ribavirin administration

At the time of randomization, subjects in Arm 2 will be initiated on the appropriate weight-based dose to be taken with food. Subjects < 75kg will be initiated on RBV 400mg enterally in the morning (QAM) and 600mg enterally at night (QPM). Subjects  $\ge 75$ kg will be initiated on RBV 600mg enterally in the morning and night (BID).

This medication will be administered predominantly outpatient, although it may be started or continued on both general hospital floors as well as the ICU.

Ribavirin dosing may be adjusted as medically required for toxicity (see section iii).

# iii. Dosage adjustment of ribavirin

| Laboratory Abnormality | Reduction in current ribavirin dose |
|---|---|
| Hgb 8.5 to <10 g/dL and/or decrease | 1. Decrease dose to 600mg daily |
| by > 2 g/dL within 4 weeks | (200mg QAM, 400mg QPM) |
| | 2. If Hgb < 12 g/dL despite 4 weeks of dose reduction in subjects with a history of stable cardiac disease, discontinue ribavirin |
| Hgb <8.5 g/dL | Discontinue ribavirin |
| WBC <1000 mm <sup>3</sup> and/or ANC <500 mm <sup>3</sup> | Discontinue ribavirin |
| Platelets < 25 k/mm <sup>3</sup> | Discontinue ribavirin |
| eGFR 30-50 ml/min | Alternating doses, 200mg and 400mg every other day |

# 5.2 Prohibited Interventions

Medications listed below will be prohibited during treatment period.

| Concomitant Drug Class: | Effect on Concentration | Clinical Comment |
|---|---|---|
| Drug Name | | |
| Antiarrhythmics: | Effect on amiodarone, ledipasvir, and | Coadministration of amiodarone |
| amiodarone | sofosbuvir concentrations unknown | with HARVONI may result in seri- |
| | | ous symptomatic bradycardia. The |
| | | mechanism of this effect is un- |
| | | known. Coadministration of amio- |
| | | darone with HARVONI is not rec- |
| | | ommended; |
| Anticonvulsants: | Decreases ledipasvir | Coadministration of HARVONI |
| carbamazepine | Decreases sofosbuvir | with carbamazepine, phenytoin, |
| phenytoin | Decreases GS-331007 | phenobarbital, or oxcarbazepine is |
| phenobarbital | | expected to decrease the concentra- |
| oxcarbazepine | | tion of ledipasvir and sofosbuvir, |
| | | leading to reduced therapeutic effect |
| | | of HARVONI. Coadministration is |
| | | not recommended. |
| Antimycobacterials: | Decreases sofosbuvir | Coadministration of HARVONI |
| Rifabutin | Decreases GS-331007 | with rifabutin or rifapentine is ex- |
| Rifampin | | pected to decrease the concentration |
| Rifapentine | | of sofosbuvir, leading to reduced |
| | | therapeutic effect of HARVONI. Coadministration is not recom- |
| | | mended mended |
| | | Coadministration of HARVONI |
| | | with rifampin, an intestinal P-gp |
| | | inducer, is not recommended |
| Herbal supplements: | Decreases sofosbuvir | Coadministration of HARVONI |
| St. John's wort (Hypericum | Decreases GS-331007 | with ST. Joh's wort, an intestinal P- |
| perforatum) | | gp inducer, is not recommended |
| HMG-CoA Reductase In- | Increases rosuvastatin | Coadministration of HARVONI |
| hibitors: | | with rosuvastatin may significantly |
| Rosuvastatin | | increase the concentration of rosu- |
| | | vastatin which is associated with |
| | | increased risk of myopathy, includ- |
| | | ing rhabdomyolysis. Coadministra- |
| | | tion of HARVONI with rosuvastat |
| | | in not recommended |

Version 6

# 5.3 Adherence Assessment

Adherence to study intervention will be assessed at all study visits noted on the Schedule of Evaluations (Section 6.1).

Subjects will have adherence assessed based on medication counts. This will be utilized in a subanalysis to determine if measured adherence rates of < 80% impact clinical outcomes in each Arm.

# 6. CLINICAL AND LABORATORY EVALUATIONS

# 6.1 Schedule of Evaluations

| | Baseline /<br>Randomi-<br>zation | | Days | | Week 1 | Week 2 | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 | Week 32 | Week 36 | End of<br>Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day Post-Randomization | 0 | <b>~</b> | 2 | 4 | 7 | 41 | 28 (+/-5 days) | 56 (+/-5 days) | 84 (+/-5 days) | 112 (+/-5 days) | | 168 (+/-5 days) | | 252 (+/-5 days) | |
| Informed Consent Obtained | X | | | | | | | | | | | | | | |
| Randomization | X | | | | | | | | | | | | | | |
| Review of Inclusion and Exclusion Criteria | Х | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | |
| Liver Transplant Recipient | Х | | | | | | | | | | | | | | |
| Liver Transplant Donor | Х | | | | | | | | | | | | | | |
| Vital Signs | Х | | | | | | 0 | 0 | 0 | 0 | | 0 | | 0 | |
| Laboratory Assessments | X | | | | | | Х | Х | Х | 0 | | 0 | | 0 | |
| Hepatitis C Viral Load Test (HCV PCR RNA) | Х | | | | | | Х | Х | Х | Х | | Х | | Х | |
| EKG | X | | | | | | | | | | | | | Χ | |
| Review of Immunosuppressants | X | | | | | | Х | Х | Х | Х | | Х | | Χ | |
| Viral Substitutions | X | | | | | | 0 | 0 | 0 | 0 | | 0 | | 0 | |
| Pregnancy Test (within 48 hrs of randomization) | Х | | | | | | | | | | | | | | |
| Review of Prohibited Medications | X | | | | | | Х | Х | Х | | | | | | |
| Study Drug Compliance | | | | | | | Χ | Χ | Χ | | | | | | |
| Virologic Failure | | | | | | | | | | | | | | | Х |
| Liver Allograft Biopsy | | | | | | | 0 | 0 | 0 | 0 | | 0 | | 0 | |
| Fibro Scan | 0 | | | | | | 0 | 0 | 0 | | | | | | |
| Adverse Events | Х | | | | | | Χ | Χ | Χ | Х | | Χ | | Χ | |
| End of Study | | | | | | | | | | | | | | | Х |

X=required; O=optional

# 6.2 Timing of Evaluations

#### 6.2.1 Pre-Randomization Evaluations

These evaluations occur prior to the subject receiving any study interventions.

# Baseline

The evaluations listed under the Baseline visit may be performed up to 14 days prior to randomization, with the exception of the pregnancy test, which must be performed within 48 hours of randomization. Additionally, HCV PCRs may be performed up to 30 days prior to randomization, provided that it was performed after the liver transplant.

Once the subject has been successfully screened and accepted for randomization, randomization must be complete within 48 hours. All subjects randomized will be included in the intent-to-treat analysis.

#### 6.2.2 Intervention and Evaluations

Once the subject has been successfully randomized, the intervention should be initiated upon that day, but must be initiated within 5 days in case of extenuating circumstances.

Study evaluations must take place within the time window indicated on the Schedule of Evaluations (Section 6.1).

#### 6.2.3 Intervention Discontinuation Evaluations

At the scheduled time of intervention discontinuation (EOT, last date of study medication), the following evaluations must be completed: HCV PCR and HCV viral substitutions (in the event of virologic failure)

If a subject prematurely terminates study intervention, a visit will be scheduled with the Principal-Investigator (PI) or designee within 72 hours to evaluate the reason for early termination. The PI or designee will attempt to resolve any issues leading to early termination and encourage the subject to resume study intervention as soon as possible. It will be clarified whether they are terminating from all components of the trial or only from the primary intervention component of the trial. If possible, the subjects will be encouraged to continue to be followed and evaluated according to the Schedule of Evaluations (Section 6.1) even if they no longer wish to receive study treatment.

Subjects that discontinue intervention due to virologic failure will be withdrawn from the study and deemed a treatment failure. These subjects may receive alternative treatment at

the investigator's discretion. SOF/LDV will be supplied upon request and RBV will be reimbursed by Gilead Sciences, Inc for up to 24 weeks if requested.

## 7. MANAGEMENT OF COMMON OR EXPECTED ADVERSE EXPERIENCES

The severity of adverse events will be determined using the grading system outlined in the NCI Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE), as it best fits the diagnostic terminology used in naming the event at the site clinical level.

# SOFOSBUVIR/LEDIPASVIR OR RIBAVIRIN (ADVERSE EVENTS IN COMMON)

| CTCAE SOC | Adverse Event | Grade Description | Criteria for<br>Modification of<br>Intervention | Procedure for Modification |
|---|---|---|---|---|
| General disor- | Fatigue | 1 – Relieved by rest | Grade 3 or if | Intervention can be withheld |
| ders and ad-<br>ministration<br>site conditions | | 2 – Not relieved by<br>rest; limiting instru-<br>mental ADL | study participant resolution, the case will discussed with the medic | for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention |
| | | 3 – Not relieved by<br>rest; limiting self-<br>care ADL | | may be discontinued. |
| Nervous system | Headache | 1 – Mild pain | Grade 3 or if | Intervention can be withheld |
| disorders | | 2 – Moderate pain;<br>limiting instrumental<br>ADL | requested by<br>study participant | for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention |
| | | 3 – Severe pain; lim-<br>iting self-care ADL | | may be discontinued. |
| Gastrointestinal disorders | Nausea | 1 – Loss of appetite<br>without alteration in<br>eating habits | Grade 3 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be |
| | | 2 – Oral intake decreased without significant weight loss, dehydration or malnutrition | | discussed with the medical monitor and the intervention may be discontinued. |
| | | 3 – Inadequate oral<br>caloric or fluid in-<br>take; tube feeding,<br>TPN, or hospitaliza-<br>tion indicated | | |
| Gastrointesti-<br>nal disorders | Vomiting | 1 – 1-2 episodes<br>(separated by 5<br>minutes) in 24 hours | Grade 3 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be |
| | | 2 – 3-5 episodes<br>(separated by 5 min)<br>in 24 hours | | discussed with the medical<br>monitor and the intervention<br>may be discontinued. |

| | | 3 - ≥ 6 episodes (separated by 5 min);<br>tube feeding, TPN or<br>hospitalization indicated | | |
|---|---|---|---|---|
| Gastrointestinal disorders | Diarrhea | 1 - Increase of < 4<br>stools per day over<br>baseline; mild in-<br>crease in ostomy<br>output compared to<br>baseline | Grade 3 if requested by study participant, treatment-resistant or recurrent; Grade 4 | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| | | 2 – Increase of 4-6<br>stools per day over<br>baseline; moderate<br>increase in ostomy<br>output compared to<br>baseline | or 5 | Grade 5: Intervention will be permanently discontinued |
| | | 3 – Increase of ≥ 7<br>stools per day over<br>baseline; inconti-<br>nence; hospitaliza-<br>tion indicated; severe<br>increase in ostomy<br>output compared to<br>baseline; limiting self<br>care ADL | | |
| | | 4 – Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated | | |
| | | 5 - Death | | |
| Psychiatric<br>disorders | Insomnia | 1 – Mild difficulty<br>falling asleep, staying<br>asleep or waking up<br>early | If requested by study participant | Intervention can be withheld<br>for up to 5 days. If there is no<br>resolution, the case will be<br>discussed with the medical |
| | | 2 – Moderate difficul-<br>ty falling asleep,<br>staying asleep or<br>waking up early | | monitor and the intervention may be discontinued. |
| | | 3 – Severe difficulty<br>in falling asleep,<br>staying asleep or<br>waking up early | | |
| Musculoskele- | Arthralgia | 1 – Mild pain | Grade 3 or if | Intervention can be withheld |
| tal and connec-<br>tive tissue dis-<br>orders | | 2 – Moderate pain;<br>limiting instrumental<br>ADL | requested by<br>study participant | for up to 5 days. If there is no<br>resolution, the case will be<br>discussed with the medical<br>monitor and the intervention |
| | | 3 – Severe pain; lim-<br>iting self care ADL | | may be discontinued. |

# 18 LIVE-C-Free

# Version 6

| Renal and urinary disorders | Chronic kidney disease | 1 - CrCl < LLN-60ml/min/1.73m2; proteinuria 2+ present; urine protein/creatinine > 0.5 2 - CrCl 59-30m/min/1.73m2 3 - CrCl 29-15ml/min/1.73m2 4 - < 15ml/min/1.73m2; dialysis indicated 5 - Death | Grade 2 | Sofosbuvir/Ledipasvir to be held if CrCl <40ml/min/1.73m2. Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Ribavirin dose should be reduced to alternating doses of 200mg and 400mg every other day if CrCl 30-50ml/min/1.73m2 Interventions can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
|---|---|---|---|---|
| Investigations | Blood bilirubin | 1 - >ULN - 1.5x ULN | Grade 3-4 | Intervention can be withheld |
| investigations | increased | 2 - >1.5-3x ULN | Grade 3-4 | for up to 5 days. If there is no |
| | | 3 - >3-10x ULN | | resolution, the case will be discussed with the medical |
| | | 4 - >10x ULN | | monitor and the intervention |
| | | | | may be discontinued. |
| Investigations | Lipase increased | 1 - > ULN-1.5x ULN | Grade 3-4 | Intervention can be withhele for up to 5 days. If there is no resolution, the case will be discussed with the medical |
| | | 2 - >1.5-2x ULN | | |
| | | 3 - >2-5x ULN | | |
| | | 4 - >5x ULN | | monitor and the intervention may be discontinued. |

# Ribavirin

| CTCAE SOC | Adverse Event | Grade Description | Criteria for<br>Modification of<br>Intervention | Procedure for Modification |
|---|---|---|---|---|
| Blood and lym-<br>phatic system | Anemia | 1 – Hgb <lln-<br>10g/dL</lln-<br> | Grade 2, modifications to dosage | Grade 2: see dosage adjustment procedure in section |
| disorders | | 2 - Hgb <10-8g/dL | Grade 3-5: per- | 5.1.iii |
| | | 3 - < 8g/dL | manently discon-<br>tinue ribavirin | Grade 3-5: ribavirin will be permanently discontinued. |
| | | 4 – Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated | | Subject experiencing Grade 3 or 4 will continue the study intervention and follow study |

| | | 5 – Death | | evaluations as detailed in section 6.1 |
|---|---|---|---|---|
| Blood and lym-<br>phatic system<br>disorders | Hemolysis | 1 – Laboratory evidence of hemolysis only (e.g. DAT, Coombs', schistocytes, decreased haptoglobin) 2 – Evidence of hemolysis and ≥ 2g/dL decrease in Hgb 3 – Transfusion or | Grade 2: modifications to dosage Grade 3-5: permanently discontinue | Grade 2: see dosage adjustment procedure in section 5.1.iii Grade 3-5: intervention will be permanently discontinued. |
| | | medical intervention indicated 4 - Life-threatening consequences; urgent intervention indicated 5 - Death | | |
| Hepatobiliary<br>disorders | Hepatic failure | 3 – Asterixis; mild<br>encephalopathy;<br>limiting self care ADL<br>4 – Moderate to se-<br>vere encephalopathy;<br>coma; life-<br>threatening conse-<br>quences<br>5 – Death | Grade 3-5 | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| Immune system<br>disorders | Allergic reaction | 1 – Transient flushing or rash, drug fever < 38 degrees C; intervention not indicated 2 – Intervention indicated; responds promptly to symptomatic treatment; prophylactic medications indicated for ≤ 24 hours | Grade 3-5 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| | | 3 – Prolonged (not<br>rapidly responsive to<br>symptomatic medica-<br>tion); recurrence of<br>symptoms following<br>initial improvement;<br>hospitalization indi-<br>cated for clinical<br>sequelae | | |

| | | 4 - Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated<br>5 - Death | | |
|---|---|---|---|---|
| Immune system disorders | Anaphylaxis | 3 – Symptomatic bronchospasm, with or without urticarial; parenteral intervention indicated; allergy-related edema/angioedema; hypotension 4 – Life-threatening consequences; urgent intervention indicated 5 – Death | Grade 3-5 | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| 0 | P | | 0 1 0 5 | 1 311 11 |
| Gastrointestinal disorders | Pancreatitis | 2 - Enzyme elevation or radiologic findings only 3 - Severe pain; vomiting; medical intervention indicated (e.g. analgesia, nutritional support) 4 - Life-threatening consequences; urgent intervention indicated 5 - Death | Grade 3-5 | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| General disor-<br>ders and ad-<br>ministration<br>site conditions | Irritability | 1 – Mild; easily consolable 2 – Moderate; limiting instrumental | Grade 3 or if<br>requested by<br>study participant | Intervention can be withheld<br>for up to 5 days. If there is no<br>resolution, the case will be<br>discussed with the medical<br>monitor and the intervention |
| | | ADL; increased attention indicated | | may be discontinued. |
| | | 3 – Severe abnormal<br>or excessive re-<br>sponse; limiting self<br>care ADL; inconsola-<br>ble | | |
| Skin and subcu-<br>taneous tissue<br>disorders | Pruritis | 1 – Mild or localized;<br>topical intervention<br>indicated | Grade 3 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be |

| | | 2 – Intense or wide- | | discussed with the medical |
|---|---|---|---|---|
| | | spread; intermittent; skin changes from scratching (e.g. edema, papulation, excoriations, lichenification, oozing/crusts); oral intervention indicated; limiting instrumental ADL 3 – Intense or widespread; constant; limiting self care ADL or sleep; oral corticosteroid or immunosuppressive therapy indicated | | monitor and the intervention may be discontinued. |
| Respiratory,<br>thoracic and<br>mediastinal<br>disorders | Dyspnea | 1 – Shortness of breath with moderate exertion 2 – Shortness of breath with minimal exertion; limiting instrumental ADL 3 – Shortness of breath at rest; limiting self care ADL 4 – Life-threatening consequences; urgent intervention indicated | Grade 3-5 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| Museulaslasla | Maralaia | 5 – Death | Grade 3 or if | |
| Musculoskele-<br>tal and connec-<br>tive tissue dis-<br>orders | Myalgia | 1 - Mild pain 2 - Moderate pain; limiting instrumental ADL 3 - Severe pain; limiting self care ADL | requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| Investigations | Neutrophil<br>count decreased | 1 - <lln-1500 -="" 1000="" 2="" 3="" 4="" <1000-500="" <1500-="" <500="" mm3="" mm3<="" td=""><td>Grade 3-4</td><td>Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued.</td></lln-1500> | Grade 3-4 | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| Psychiatric<br>disorders | Depression | 1 – Mild depressive<br>symptoms<br>2 – Moderate depres-<br>sive symptoms; limit-<br>ing instrumental ADL | Grade 3-5 or if<br>requested by<br>study participant | Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention |

| 3 – Severe<br>symptoms;<br>self care Al<br>talization r<br>cated | DL; hospi- | may be discontinued. Grade 5: Intervention will be permanently discontinued |
|---|---|---|
| 4 - Life-thr<br>consequen<br>threats of h<br>self or othe<br>talization i | ces;<br>narm to<br>ers; hospi- | |
| 5 – Death | | |

# Transplant and Immunosuppression-related

| CTCAE SOC | Adverse Event | Grade Description | Criteria for<br>Modification of<br>Intervention | Procedure for Modification |
|---|---|---|---|---|
| Infections and infestations | Abdominal infection | 3 – IV antibiotic,<br>antifungal, or antivi-<br>ral intervention indi-<br>cate; radiologic or<br>operative interven-<br>tion indicated | Grade 4-5 | Grade 4: Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| | | 4 – Life-threatening consequences; urgent intervention indicated 5 – Death | | Grade 5: Intervention will be permanently discontinued |
| Infections and infestations | Biliary tract<br>infection | 3 – IV antibiotic,<br>antifungal, or antivi-<br>ral intervention indi-<br>cate; radiologic or<br>operative interven-<br>tion indicated | Grade 4-5 | Grade 4: Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| | | 4 – Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated | | Grade 5: Intervention will be permanently discontinued |
| | | 5 – Death | | |
| Infections and infestations | Hepatic infection | 3 – IV antibiotic,<br>antifungal, or antivi-<br>ral intervention indi-<br>cate; radiologic or<br>operative interven-<br>tion indicated | Grade 4-5 | Grade 4: Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. |
| | | 4 - Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated | | Grade 5: Intervention will be permanently discontinued |
| | | 5 – Death | | |

| T. C | CMW | 1 Indus COM | C 1. 4.5 | Cond. A John Co. |
|---|---|---|---|---|
| Infections and infestations | CMV | 1 – Isolation of CMV<br>from blood or sterile<br>site or positive CMV<br>PCR without clinical<br>symptoms | Grade 4-5 | Grade 4: Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| | | 2 – Isolation of CMV from blood or sterile site or positive CMV PCR with clinical symptoms (fever, malaise, leukopenia, thrombocytopenia) 3 - Isolation of CMV from blood or sterile site or positive CMV PCR with clinical symptoms (fever, malaise, leukopenia, thrombocytopenia) and histological evidence of viral cytopathic effect or positive CMV culture from a deep tissue specimen 4 - Life-threatening | | |
| | | consequences; ur-<br>gent intervention<br>indicated | | |
| | | 5 – Death | | |
| Infections and infestations | Wound infection | 2 – localized; local<br>intervention indicat-<br>ed (e.g. topical anti-<br>biotic, antifungal,<br>antiviral) | Grade 4-5 | Grade 4: Intervention can be withheld for up to 5 days. If there is no resolution, the case will be discussed with the medical monitor and the intervention may be discontinued. Grade 5: Intervention will be permanently discontinued |
| | | 3 – IV antibiotic,<br>antifungal, or antivi-<br>ral intervention indi-<br>cated; radiologic or<br>operative interven-<br>tion indicated | | |
| | | 4 - Life-threatening<br>consequences; ur-<br>gent intervention<br>indicated 6 - Death | | |
| | | o - Death | | |

# 8. CRITERIA FOR INTERVENTION DISCONTINUATION

The intervention will be withheld/discontinued for specific grades of adverse effects as detailed in section 7. Additionally, the intervention will be discontinued if the subject meets criteria for the following reasons:

Virologic failure, defined as:

<u>Breakthrough</u>: HCV RNA  $\geq$  LLOQ after having previously had HCV RNA  $\leq$  LLOQ, while on treatment, confirmed with 2 consecutive values (note: second confirmation value can be posttreatment), or last available on-treatment measurement with no subsequent follow up values, OR

<u>Rebound</u>: > 1 log10IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (note: second confirmation value can be post-treatment), or last available on-treatment measurement with no subsequent follow up values, OR

Nonresponse: HCV RNA persistently  $\geq$  LLOQ through 8 weeks of treatment, OR Relapse: HCV RNA  $\geq$  LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement

Pregnancy: If a woman becomes pregnant or a male's female partner becomes pregnant while on-study, the subject will be required to instruct investigators immediately. If he/she is in Arm 1, he/she may remain on therapy but will be ineligible for treatment with ribavirin in the event of virologic failure. If he/she is in Arm 2, therapy must be discontinued immediately and the subject will be counseled on the potential risks of exposure by the PI or designee. A discussion will occur with the medical monitor to decide whether the subject is eligible to be continued on sofosbuvir/ledipasvir alone.

Loss of graft: Defined as death or need for retransplant. Patients will be deemed a treatment failure and the intervention will be discontinued.

### 9. STATISTICAL CONSIDERATIONS

### 9.1 General Design Issues

This is a multi-center, prospective, randomized, open-label, intent-to-treat pilot study.

The primary objective is to estimate the effect that LDV/SOF for 12 weeks will have on SVR12 compared to LDV/SOF plus ribavirin for 12 weeks.

Version 6

#### 9.2 Outcomes

- 9.2.1 Primary outcome Treatment efficacy, defined as the proportion of subjects achieving sustained virologic response 12 (SVR12) weeks after completing the antiviral regimen
- 9.2.2 Secondary outcomes Secondary endpoints include the proportion of subjects achieving clearance of viremia during therapy, at the end of therapy, week 4 and 24 SVR (week 4, week 8, EOT, SVR4, SVR24).
- 9.2.3 Safety outcomes Overall safety and tolerability of each regimen will be estimated by measuring the incidence of adverse drug reactions and the development of medication intolerance requiring dose reduction, temporary withdrawal, or removal of the study drug(s), incidence of the need for supportive medications (erythropoietins, colonystimulating factors), incidence of intolerance requiring dose reduction, temporary withdrawal, or removal of immunosuppressants, overall and opportunistic infections, biopsyproven rejection rates, death, and graft loss. Other safety outcomes include virologic mutations based on NS5A and NS5B viral substitutions at baseline and in the event of virologic failure.

# 9.3 Sample Size Estimation for the Primary Outcome

For a definitive trial, if we assume an efficacy rate of 95% with an acceptable noninferiority margin of 10%, 75 subjects would be needed in each arm to provide an alpha level of 0.05 with 80% power to demonstrate noninferiority. Assuming a 10% dropout rate (indicating randomization, but failure to receive a dose of study medication), 85 subjects would need to be randomized in each arm. In this pilot study of 50 subjects, we will be able to obtain estimates of these rates for the two groups for use in the future definitive trial.

# 9.4 Statistical Evaluation of Primary Endpoint

# 9.4.1 Statistical Hypotheses:

The specific null and alternative hypotheses for comparing these two treatments in a non-inferiority design are:  $H_0$ :  $\pi_{LDV/SOF+ribavirin} - \pi_{LDV/SOF} = \delta_o$  and  $H_A$ :  $\pi_{LDV/SOF+ribavirin} - \pi_{LDV/SOF} < \delta_o$  (non-inferior) where  $\delta_o$  =0.10. where  $\pi_{LDV/SOF+ribavirin}$  (assumed to be 95%) represents the proportion with a successful outcome due to treatment with LDV/SOF plus ribavirin for 12 weeks and  $\pi_{LDV/SOF}$  represents the proportion of a successful outcome due to treatment with LDV/SOF for 12 weeks.

# 9.4.2 Efficacy Analysis:

Although there is insufficient power to conduct any formal statistical analyses, preliminary estimates of effects for treatment comprisons will be intent-to-treat, where all randomized subjects will be included in the analysis and each subject will be included in the treatment to which they were randomized.

Baseline demographics and clinical outcomes will be presented by treatment. Estimates of the differences between these, along with 95% confidence intervals, will be generated. The primary outcome of proportion of subjects with success (defined as the proportion of subjects achieving sustained virologic response 12 (SVR12) weeks after completing the antiviral regimen) as well as estimates of all secondary outcomes for each treatment will be reported along with 95% confidence intervals.

### 9.7 Safety Analysis

## 9.7.1 Safety Outcomes

Safety outcomes include the proportion of subjects who experience any treatment-related serious adverse events (SAEs) during the treatment phase and up to 30 days following completion of the treatment.

Overall safety and tolerability of each regimen will be estimated by measuring the incidence of:

- Development of medication intolerance requiring dose reduction, temporary withdrawal, or removal of the study drug(s)
- Incidence of the need for supportive medications (erythropoietins, colony-stimulating factors)
- Incidence of intolerance requiring dose reduction, temporary withdrawal, or removal of immunosuppressants
- Overall and opportunistic infections
- Biopsy-proven rejection rates
- Mortality
- Graft loss

Other specific SAEs to be monitored may be added in consultation with the DSMB. The cumulative incidences of each outcome will be estimated along with 95% confidence intervals

# 9.7.2 Interim Safety Monitoring

The Data Safety Monitoring Board (DSMB) will review study safety event rates, center performance, adverse events (AEs), and serious adverse events (SAEs) periodically. This review will identify any clinical, operational, or other data issues that might require changes or adjustments in the way in which the trial is conducted as well as any safety issues that may need to be addressed. In order to accommodate this, the Data Coordination Unit (DCU) will generate safety monitoring reports as well as a comprehensive statistical report periodically for the DSMB. These reports will contain compiled data on enrollment, demographic and baseline characteristics, eligibility and protocol violations, safety data, concomitant medications and procedures, and data quality (e.g., timeliness of data entry, and number of data clarification requests generated and resolved). All AEs and SAEs will be coded using MedDRA and summarized in terms of frequency of the event, number of subjects having the event, timing relative to randomization, and severity and relatedness to treatment. For each review, the DCU will generate two statistical reports – an open, blinded report to be distributed to the Executive Committee and the DSMB, and a closed report to be distributed only to the DSMB. For the closed report only, the statistics will also be provided by partially blinded treatment group (A vs B). If the DSMB wishes to be completely unblinded for closed reports, a sealed treatment identification envelope will be provided to the DSMB; this envelope can be opened at the discretion of the DSMB. The closed report will also contain data listings identifying subjects with specific safety outcomes such as mortality.

## 9.7.3 Stopping the Trial Based on Interim Safety Data

In case of concern for safety issue arises from DSMB, the trial may be stopped temporarily or permanently if the serious adverse event rate (SAEs related to the study treatment) exceeds a clinically acceptable rate of 10% in either arm. Data for events will not be evaluated until the first 30 subjects have completed 30 day post treatment follow-up for each arm.

## 10. DATA COLLECTION, SITE MONITORING, ADVERSE EVENT REPORTING

### 10.1 Data Processing

Data management will be handled by DCU. All study activities will be conducted in coordination with the study PI, and will use an electronic data acquisition method where all clinical data on enrolled subjects will be entered by the site personnel in real time. The latest version of each CRF will be available as a PDF file on the study website for

use as worksheets and source documents by study personnel. The study data will be managed (including data queries) by DCU using the WebDCU<sup>TM</sup> system. This user-friendly web-based database system, developed by DCU, will be used for regulatory document management, subject randomization, data entry, data validation, project progress monitoring, subject tracking, user customizable report generation and secure data transfer.

## 10.2 Data Security and Confidentiality

During the course of the trial, user access to the files with subject identifiers, treatment assignment and files with study outcomes will be restricted to core staff. In addition to use of passwords and other security measures, all documents containing identifying information on individuals or physicians are considered confidential materials and will be safeguarded to the greatest possible extent. No information, which identifies a specific person, hospital, or physician, will be released to, or discussed with anyone other than study team members.

Because the DCU uses a web-based system, source documents and CRFs will remain at the participating sites. The study database only identifies study subjects by unique study identification codes. All data will be stored in a manner that is HIPAA compliant, without the ability to track the information back to a specific subject except through a password protected system. All collected information about a subject will be stored by a unique identification code. All DCU personnel have current Human Subjects Protection Training Certification. Clinical information will not be released without written permission of the subject, except as necessary for monitoring by IRB, the FDA, OHRP, the sponsor, or the sponsor's designee.

### 10.3 Data Quality Assurance

The study data will be managed (including data queries) by DCU using the WebDCU<sup>TM</sup> system. This user-friendly web-based database system, developed and validated by the DCU, will be used for regulatory document management, subject randomization, data entry, data validation, project progress monitoring, subject tracking, user customizable report generation and secure data transfer. In addition to the study database, the DCU will provide the clinical site staff access (via password) to a standard set of web-enabled tools, including subject visit calendar, subject accrual status, case report form completion status, and outstanding data clarification request status pertaining to their respective clinical sites. Furthermore, all approved study materials, such as the protocol, informed consent template and manual of procedures, will be housed on the website to ensure that the clinical sites always have access to the most current trial documents.

Data should be independently entered by the designated personnel at each clinical site into WebDCU<sup>TM</sup> within the time intervals specified in the schedule of assessments. Enrollment data, however, must be entered into the WebDCU<sup>TM</sup> database before the subject can be randomized. Serious adverse events must be entered into the WebDCU<sup>TM</sup> within 24 hours of the site staff's first awareness of the event. It is critically important to the effective and efficient conduct of the study that data be entered in a timely manner. An electronic copy of the CRFs will be made available to the clinical sites prior to initiation of the study to be used as worksheets to capture the required data for the study. The DCU staff will perform range verification, consistency checks, and quality assurance on the data. The staff at the DCU will contact the sites regarding missing data or queries on CRF data. They will maintain direct contact with the staff at the participating sites to ensure the study is conducted according to the Good Clinical Practice Guidelines and all applicable regulations.

Experienced clinical research monitors will be contracted through the DCU to perform on site source data verification (SDV) of key outcome and safety data variables during the study. In addition to data verification, the monitor will evaluate drug accountability and site facilities. The CRFs and corresponding source documents should be made available to the study monitor at each site visit. It is also expected that the PI, or a designated member of the research staff, will be available during the monitoring visit to review the data and resolve any queries.

## 10.4 Adverse Experience Reporting

In order to ensure prompt reporting of adverse events, all adverse events (as well as all related study data) must be entered into the WebDCU<sup>TM</sup> within five days of collection date. All serious adverse events (SAEs) must be reported on the WebDCU<sup>TM</sup> within 24 hours of the study site staff first being made aware of its occurrence. The site investigators are required to provide relevant information, including description of the adverse event, date/time of onset and resolution, severity and seriousness, action taken, and suspected relationship to the study treatment.

Reporting of any serious adverse event will trigger notification of the event to the DCU Project Manager (PM) and the independent Medical Safety Monitor (MSM). The MSM will conduct an independent review of each of these events to determine if it is serious, unexpected, and study treatment related.

Periodically throughout the study, the MSM will review reports on the incidence rates of all reported adverse events, whether serious or not. Should such monitoring uncover issues that may threaten subject safety (e.g. unexpectedly high rate of adverse events), the study statistician and principal investigator will prepare a report to be submitted to the DSMB for their review and further actions to be taken, if any.

#### 11. HUMAN SUBJECTS

# 11.1 Institutional Review Board (IRB) Review and Informed Consent

This protocol, the ICF, and any subsequent modifications must be reviewed and approved by the local IRB at each of the participating institutions. A signed and dated ICF must be obtained from the subject as defined in 21CFR50.3. The ICF must also be signed and dated by a member of the study staff qualified to be delegated the authority to obtain informed consent, and a witness (if required by the local IRB). A copy of the ICF must be given to the subject and the consent process must be documented in the subject's medical record. The PI or delegated sub-Investigator is responsible for ensuring that informed consent is obtained from each patient prior to conducting any study-related activities.

No deviations from or changes to the study protocol should be initiated except when necessary to eliminate immediate hazard to the subject. However, the IRB, DCU, and Study Sponsor must be informed of this as soon as possible thereafter. It is the study site PI's responsibility to report SAEs occurring during the study to their IRB, as required and as soon as possible.

# 11.2 Study Modification/Discontinuation

The study may be modified or discontinued at any time by the IRB, the sponsor, the OHRP, the FDA, or other government agencies as part of their duties to ensure that research subjects are protected.

## 12. PUBLICATION OF RESEARCH FINDINGS

Publication of the results of this trial will be reviewed and approved by all coinvestigators. Final results will be submitted to ClinicalTrials.gov. Any presentation, abstract, or manuscript will be made available for review by the sponsor prior to submission.

#### 13. REFERENCES

- 1. Gordon FD, Kwo P, Ghalib R. Peginterferon alfa-2b and ribavirin for hepatitis C recurrence post orthotopic liver transplantation. J Clin Gastroenterol. 2012; 46: 700-708.
- 2. Gane EJ, Stedman CA, Hyland RH, et.al. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med. 2013; 368(1): 34-44.
- 3. Lawitz E, Mangia A, Wyles D, et.al. Sofosbuvir for previously untreated hepatitis C infection. N Engl J Med. 2013; 368(20): 1878-87.
- 4. Lawitz E, Poordad FF, Pang PS, et.al. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naïve and previously treated patients with genotype 1 hepatitis C infection (LONESTAR): an open-label, randomized, phase 2 trial. Lancet. 2014; 383(9916): 515-23.
- 5. OPTN/SRTR Annual Data Report: Liver. Am J Transplant. 2014; 14(S1): 69-96.
- 6. Charlton M, Gane E, Manns M, et.al. Sofosbuvir and RBV for the treatment of established recurrent HCV infection after liver transplantation: preliminary results of a prospective, multicenter study. Hepatology. 2013; 58: LB2.
- 7. Bzowej N, Nelson D, Terrault D, et.al. PHOENIX: a randomized controlled trial of peginterferon alfa-2a plus ribavirin as a prophylactic treatment after liver transplantation for hepatitis C virus. Liver Transpl. 2011; 17: 528-38.
- 8. Curry MP, Forns X, Chung RT, et.al. Pretransplant sofosbuvir and ribavirin to prevent recurrence of HCV infection after liver transplant. Hepatology. 2013; 58(S4): 314A-5A.
- 9. Guedj J, Pang PS, Denning J, et.al. Analysis of hepatitis C viral kinetics during administration of two nucleotide analogues: sofosbuvir (GS-7977) and GS-0938. Antivir Ther. 2014; 19(2): 211-20.
- 10. Powers KA, Ribeiro RM, Patel K, et.al. Kinetics of hepatitis C virus reinfection after liver transplantation. Liver Transpl. 2006; 12(2): 207-16.

#### APPENDIX I

US Public Health Service (PHS)Guideline for Reducing Human Immunodeficiency Virus, Hepatitis B Virus, and Hepatitis C Virus Transmission Through Organ Transplantation, 2013 ed.

Donor at Increased Risk for recent HIV, HBV, and HCV infection

- 1. People who have had sex with a person known or suspected to have HIV, HBV, or HCV infection in the preceding 12 months
- 2. Men who have had sex with men (MSM) in the preceding 12 months
- 3. Women who have had sex with a man with a history of MSM behavior in the preceding 12 months
- 4. People who have had sex in exchange for money or drugs in the preceding 12 months
- 5. People who have had sex with a person who had sex in exchange for money or drugs in the preceding 12 months
- 6. A child who is  $\leq$  18 months of age and born to a mother known to be infected with, or at increased risk for, HIV, HBV, or HCV infection
- 7. A child who has been breastfed within the preceding 12 months and the mother is known to be infected with, or at increased risk for, HIV infection
- 8. People who have injected drugs by intravenous, intramuscular, or subcutaneous route for non-medical reasons in the preceding 12 months
- 9. People who have been in lockup, jail, prison, or a juvenile correctional facility for more than 72 consecutive hours in the preceding 12 months
- 10. People who have been newly diagnosed with, or have been treated for, syphilis, gonorrhea, *Chlamydia*, or genital ulcers in the preceding 12 months
- 11. Donor who is at increased risk for recent HCV infection only:
  - a. People who have been on hemodialysis in the preceding 12 months

Version 6

# APPENDIX II Milan Criteria

- 1. A single HCC nodule with a maximum size of 5 cm OR
- 2. Up to 3 HCC nodules with the largest not exceeding 3 cm AND

No macrovascular invasion